CLINICAL TRIAL: NCT02266004
Title: Transcranial Direct Current Stimulation for Freezing of Gait in Patients With Parkinson's Disease
Brief Title: Transcranial Direct Current Stimulation for Freezing of Gait
Acronym: TDCS-FOG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult to recruit participants
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Corneliu C Luca, Assisstant Professor of Neurology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140127
Record Dates: First submitted 2014-10-07; First posted 2014-10-16 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Parkinson's Disease
Keywords: transcranial direct current stimulation; neuromodulation
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- tDCS+ LT (Experimental): Transcranial direct current stimulation(tDCS) plus locomotor training (LT) 3x per week for 3 consecutive weeks.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Other: locomotor training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Anodal tDCS will be applied for the duration of the walking training at 2 milliamps with IOMED Phoresor.
  Other Names: tDCS
Other: locomotor training — An individualized dual-task walking program for approximately 30 minutes.

SUMMARY:
This study will evaluate the effects of transcranial direct current stimulation (tDCS) in combination with locomotor training in patients with Parkinson's disease (PD) and freezing of gait (FOG).

ELIGIBILITY:
Inclusion Criteria:

1. age 18- 80
2. Parkinson's disease stages 2-3 Hoehn and Yahr.
3. Presence of Freezing of Gait
4. Stable medication regimen
5. Time to complete TUG >12 seconds

Exclusion Criteria:

1. medical condition that would interfere with walking and training for 30 minutes
2. unable to perform timed up and go in the off condition
3. history of seizures
4. implanted deep brain stimulator, pacemaker or any other electronic device.
5. dementia
6. Adults unable to consent, individuals who are not yet adults (infants, children, teenagers) pregnant women, prisoners will not be considered for participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corneliu Luca, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was removed from the study and re-enrolled. However, this participant did not complete the study intervention on their first or second enrollment. Therefore their data has not been included in any of the outcome measures.
Period: Overall Study
Arm/Group | tDCS+ LT
Started | 9
Completed | 7
Not Completed | 2
Not completed — unrelated adverse event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Walking Speed
Description: walking speed will be measured using sensors during a 90 second walk
Time Frame: baseline, 3 weeks
Population: Unable to retrieve collected data on the other 5 participants who completed the study due to a malfunction in the sensors.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 2
m/s | 0.169 (0.244)

2. Secondary Outcome: Change in Motor Scores as Measured by Unified Parkinson's Disease Rating Scale (UPDRS)
Description: UPDRS motor score range from 0-56 with higher scores indicating greater impairment.
Time Frame: baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 7
score on a scale | -1.714 (14.088)

3. Secondary Outcome: Change in Stride Length
Description: Stride length is measured with mobile sensors attached to participant's extremities during the 90 second walk.
Time Frame: baseline, 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 2
m | 0.127 (0.239)

4. Secondary Outcome: Change in Postural Sway
Description: Postural sway is measured with mobile sensors attached to participant's extremities during the 30 seconds of quiet standing.
Time Frame: baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: m^2/s^5
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 7
m^2/s^5 | -0.012 (0.009)

5. Secondary Outcome: Change in Timed Up-and-Go (TUG) Time
Description: Participants are timed while standing up from a chair, walking around a cone, and returning to their chair.
Time Frame: baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 7
seconds | -6.878 (4.268)

6. Secondary Outcome: Change in Motor Threshold
Description: Transcranial magnetic stimulation is used to measure motor threshold of the primary motor area. The motor threshold was defined as the minimum intensity needed to evoke 5 out 10 motor evoked potentials in the first dorsal interosseous muscle in the hand.
Time Frame: baseline, 3 weeks
Population: 3-week data not collected for 5 participants who completed the study.
Measure: Mean (Standard Deviation); unit: percentage of TMS output
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 2
percentage of TMS output | -0.005 (0.021)

7. Secondary Outcome: Change in Glutamate/Gamma Aminobutyric Acid(GABA) Ratio
Description: Glutamate/GABA ratio will be measured with magnetic Resonance Spectroscopy (MRS).
Time Frame: baseline, 3 weeks
Population: No data was collected for this outcome measure.
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Backward Digit Span
Description: Digit span is measured by total number of correct digits recited.
Time Frame: baseline, 3 weeks
Population: No data was collected for this outcome measure.
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in the Trail Making Test Time
Description: Trail making test is measured as the number of seconds required to complete the task, with higher scores indicating greater impairment.
Time Frame: baseline, 3 weeks
Population: No data was collected for this outcome measure.
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in the Montreal Cognitive Assessment (MOCA)
Description: The MOCA has a total score ranging from 0-30 with a higher score indicating better performance.
Time Frame: baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 7
score on a scale | 2.57 (1.89)

11. Secondary Outcome: Change in the Auditory Consonant Trigrams Test (ACT)
Description: The ACT has a score from 0-60 with higher score indicating better performance.
Time Frame: baseline, 3 weeks
Population: No data was collected for this outcome measure.
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in the Freezing of Gait Questionnaire (FOG-Q)
Description: The FOG-Q has a total score ranging from 0-24 with higher scores indicating more incidents of freezing.
Time Frame: baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS+ LT
Number analyzed (Participants) | 7
score on a scale | -4.29 (3.21)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | tDCS+ LT
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS+ LT (N=9)
dizziness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS+ LT (N=9)
fall at home (Musculoskeletal and connective tissue disorders) | 1 (2)
fatigue (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Data was not collected on 4 of the outcome measures due to lack of funding which contributed to the difficulty in performing the tests required per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT02266004/Prot_SAP_000.pdf